CLINICAL TRIAL: NCT01683058
Title: A 26-week, Multicenter, Open-label, Extension Study of Aripiprazole Intramuscular Depot (OPC-14597, Lu AF41155) in Patients With Schizophrenia
Brief Title: Open-label, Extension Study of Aripiprazole Intramuscular Depot (OPC-14597, Lu AF41155) in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry); Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-12-297
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole IM Depot (Experimental): Aripiprazole IM Depot 400 mg or 300 mg once monthly (every 28 days) for 24 weeks
  Interventions: Drug: Aripiprazole IM Depot

INTERVENTIONS:
Drug: Aripiprazole IM Depot — Aripiprazole IM Depot 400 mg or 300 mg

SUMMARY:
The phase 3 Trial 31-12-291 is part of the aripiprazole IM depot clinical development program and has been designed to demonstrate the efficacy and safety of aripiprazole IM depot for the treatment of adults experiencing an acute relapse of schizophrenia. Subjects receive treatment during a 12-week double-blind acute treatment phase. The current trial (31-12-297) will allow the subjects who complete Trial 291 to enter this open label trial at the investigator's discretion, where additional safety and tolerability data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 to 66 years of age, inclusive, at the time of informed consent.
* Subjects who are able to provide written informed consent (as required by IRB/IEC) prior to the initiation of any protocol-required procedures.
* Ability, in the opinion of the investigator, to understand the nature of the trial and follow protocol requirements, including the prescribed dosage regimens, tablet ingestion, and discontinuation of prohibited concomitant medication, and to be reliably rated on assessment scales.
* Subjects who have met the completion criteria in the 31-12-291 registrational trial for the acute treatment of adults with schizophrenia
* Subjects who, in the investigator's judgment, require chronic treatment with antipsychotic medication and would benefit from extended treatment with an IM depot formulation.
* Outpatient status at the Week 12 in Trial 291, with the exception of those subjects eligible to enter Trial 297 due to a positive interim analysis.

Exclusion Criteria:

* Sexually active males of childbearing potential who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 180 days after the last dose of trial medication. Sexually active Women of Childbearing Potential who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 150 days after the last dose of trial medication.
* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving IMP in this trial.
* Subjects experiencing acute depressive symptoms within the past 30 days, according to the investigator's opinion, that requires treatment with an antidepressant.
* Subjects who are anticipated needing CYP2D6 or CYP3A4 inhibitors or CYP3A4 inducers during the course of the trial.
* Subjects with a significant risk of violent behavior; who represent a risk of committing suicide; or who in the clinical judgment of the investigator present a serious risk of suicide.
* Subjects requiring any antipsychotic(s) other than aripiprazole IM depot after completion of Trial 291.
* Subjects likely to require prohibited concomitant therapy during the trial
* Laboratory test and ECG results which are exclusionary
* Any subject who, in the opinion of the investigator or medical monitor, should not participate in the trial

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (29):
  - Little Rock, Arkansas
  - Springdale, Arkansas
  - Carson, California
  - Escondido, California
  - Garden Grove, California
  - Long Beach, California
  - National City, California
  - Oakland, California
  - Pico Rivera, California
  - San Diego, California
  - Santa Ana, California
  - Sherman Oaks, California
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Kissimmee, Florida
  - North Miami, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Hoffman Estates, Illinois
  - Lake Charles, Louisiana
  - Flowood, Mississippi
  - St Louis, Missouri
  - Marlton, New Jersey
  - Holliswood, New York
  - Dayton, Ohio
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
- Croatia (2):
  - Popovača
  - Zagreb
- Daugavpils, Latvia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multicenter, open-label, single-arm rollover trial designed to demonstrate the safety of aripiprazole intramuscular (IM) depot [400 or 300 milligrams (mg)] for the acute treatment of participants with schizophrenia, who met completion criteria in the registration trial NCT01663532. 74 participants were enrolled in this trial.
Pre-assignment Details: Participants entered this trial after completing the Week 12/Early Termination (ET) visit of trial NCT01663532 as it served as the Baseline evaluations for this trial.
Groups:
- Aripiprazole IM Depot 400/300 mg: All participants in this trial received aripiprazole IM depot 400/300 mg every 4 weeks for over 24 weeks.
Period: Overall Study
Arm/Group | Aripiprazole IM Depot 400/300 mg
Started | 74
Completed | 45
Not Completed | 29
Not completed — Lost to Follow-up | 9
Not completed — Adverse Event | 6
Not completed — Subject Met Withdrawal Criteria | 5
Not completed — Withdrawal by Subject | 7
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Aripiprazole IM Depot 400/300 mg
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Treatment Emergent Adverse Events (TEAEs), Severe TEAEs, Discontinued Investigational Medicinal Product (IMP) Due to AEs, Serious TEAEs and Outcome of Death
Description: A TEAE was defined as an AE that began after the first injection or was continuous from Baseline and was serious, study drug-related, or resulted in death.
Time Frame: Baseline to Week 24
Population: In safety analysis, all enrolled participants took at least one injection of aripiprazole IM depot 400/300mg in the IM depot treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Aripiprazole IM Depot 400/300 mg
Number analyzed (Participants) | 74
Percentage of participants
  Participants with TEAEs | 66.2
  Participants with serious TEAEs | 6.8
  Participants with severe TEAEs | 8.1
  Participants discontinued IMP due to AEs | 8.1
  Deaths | 0.0

2. Secondary Outcome: Mean Change From Baseline in Suicidal Ideation Intensity Total Score by the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Data collected from C-SSRS were mapped into C-CASA. The Columbia Classification Algorithm of Suicide Assessment (C-CASA) method and C-SSRS(text in parentheses as said below) were mapped as; 1= completed suicide(completed suicide); 2= suicide attempt(actual attempt); 3= preparatory actions toward imminent suicidal behavior (interrupted attempt, aborted attempt and preparatory acts/behavior); 4= suicidal ideation(wish to die,active suicidal thought, active suicidal thought with method, active suicidal thought with intent,active suicidal thought with plan/intent); 5= self-injurious behavior, intent unknown; 6= not enough information: death; 7= non-suicidal self-injurious behavior(nonsuicidal self-injurious behavior); 8= other accident; psychiatric/medical; 9= not enough information/non-death. C-CASA category 5, 6, 8 and 9 are not applicable. For each item, each participant received an intensity score from 0(none) to 5(worst). Suicidal ideation intensity total score range from 0 to 25.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400/300 mg
Number analyzed (Participants) | 74
Units on a scale
  Week 4 (N= 69) | -0.1 (2.3)
  Week 8 (N= 61) | -0.1 (2.2)
  Week 12 (N= 57) | -0.3 (2.0)
  Week 16 (N= 52) | 0.7 (4.7)
  Week 20 (N= 44) | 0.3 (2.0)
  Week 24 (N= 45) | 0.0 (0.0)
  Last Visit (N= 71) | 0.6 (4.2)

3. Secondary Outcome: Mean Change From Baseline by Week by Extrapyramidal Symptoms (EPS) Evaluated Using the Simpson-Angus Scale (SAS)
Description: The EPS rating scales included SAS total score (range 10-50) was the sum of the rating scores for 10 items from the SAS panel. This scale consists of a list of 10 symptoms, each to be rated on a 5-point scale of severity. For each symptom, the rating which best described the patient's condition were, 1= gait; 2= arm dropping; 3= shoulder shaking; 4= elbow rigidity; 5= wrist rigidity; 6= head rotation; 8= tremor; 9= salivation; 10= akathisia.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400/300 mg
Number analyzed (Participants) | 72
Units on a scale
  Week 12 (N= 66) | 0.19 (1.51)
  Week 24 (N= 70) | 0.04 (1.62)

4. Secondary Outcome: Mean Change From Baseline by Week by EPS Evaluated Using the Abnormal Involuntary Movement Scale (AIMS)
Description: EPS rating scale included the AIMS movement rating score (range 0-28) was the sum of the rating scores for facial and oral movements (i.e., item 1 - 4), extremity movements (i.e. item 5 - 6), and trunk movements (i.e. item 7). The symptoms for facial and oral movements were 1= muscles of facial expression, 2= lips and perioral area, 3= jaw and 4=tongue; extremity movements were, 5= upper (arms, wrists, hands, fingers), lower (legs, knees, ankles, toes), 7= neck, shoulders, hips). This scale consisted of 10 items, each to be rated on a 4-point scale of severity, and 2 questions to be answered by yes or no. To complete the scale, the patient was observed unobtrusively at rest (e.g., in waiting room). The chair used for this examination was hard, firm one without arms.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400/300 mg
Number analyzed (Participants) | 73
Units on a scale
  Week 12 (N= 65) | -0.06 (0.81)
  Week 24 (N= 70) | 0.07 (1.28)

5. Secondary Outcome: Mean Change From Baseline by Week by EPS Evaluated Using Barnes Akathisia Rating Scale (BARS)
Description: The BARS global score (range 0-5) was derived from the global clinical assessment of akathisia from the BARS panel were, 0= absent; 1= questionable; 2= mild akathisia; 3= moderate akathisia; 4= marked akathisia; 5= severe akathisia. Patients were observed while they were seated and then standing (for a minimum of 2 minutes in each position). Symptoms were observed in other situations (e.g., while engaged in neutral conversation, engaged in activity on the ward) was also rated.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400/300 mg
Number analyzed (Participants) | 73
Units on a scale
  Week 12 (N= 65) | 0.19 (0.73)
  Week 24 (N= 70) | 0.14 (0.91)

6. Secondary Outcome: Mean Change in Body Temperature From Baseline in All Participants.
Description: The body temperature, which is a vital sign parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of treatment-emergent adverse events of potential clinical relevance included abnormal values in body temperature, heart rate, systolic and diastolic blood pressure, and respiratory rate that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: Safety sample was analyzed. All enrolled participants who took at least one injection of study medication in the IM depot treatment period. Last visit was defined as the last assessment visit in the treatment phase (scheduled or unscheduled visit).
Measure: Mean (Standard Deviation); unit: °C
Groups:
- Aripiprazole IM Depot 400/ 300 mg: All participants in this trial received aripiprazole IM depot 400/300 mg every 4 weeks for over 24 weeks.
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
°C
  Week 4 (N= 69) | 0.1 (0.4)
  Week 8 (N= 61) | -0.0 (0.4)
  Week 12 (N= 58) | 0.0 (0.4)
  Week 16 (N= 53) | 0.0 (0.3)
  Week 20 (N= 44) | 0.1 (0.4)
  Week 24 (N= 45) | 0.1 (0.4)
  Last visit (N= 72) | 0.0 (0.4)

7. Secondary Outcome: Mean Change in Heart Rate Supine From Baseline in All Participants.
Description: The heart rate supine, which is a vital sign parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of treatment-emergent adverse events of potential clinical relevance included abnormal values in body temperature, heart rate, systolic and diastolic blood pressure, and respiratory rate that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
beats/min
  Week 4 (N= 69) | 3.8 (10.9)
  Week 8 (N= 61) | 2.3 (11.2)
  Week 12 (N= 58) | 1.3 (10.8)
  Week 16 (N= 53) | 4.7 (12.0)
  Week 20 (N= 44) | 3.6 (9.8)
  Week 24 (N= 45) | 1.7 (12.7)
  Last visit (N= 72) | 3.4 (12.1)

8. Secondary Outcome: Mean Change in Systolic Supine Blood Pressure (BP) From Baseline in All Participants.
Description: The systolic supine BP, which is a vital sign parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of treatment-emergent adverse events of potential clinical relevance included abnormal values in body temperature, heart rate, systolic and diastolic blood pressure, and respiratory rate that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
mmHg
  Week 4 (N= 69) | 1.9 (12.8)
  Week 8 (N= 61) | 1.3 (12.2)
  Week 12 (N= 58) | -0.2 (12.4)
  Week 16 (N= 53) | 2.0 (12.4)
  Week 20 (N= 44) | 4.8 (12.8)
  Week 24 (N= 45) | 0.7 (11.3)
  Last visit (N= 72) | 0.4 (13.1)

9. Secondary Outcome: Mean Change in Diastolic Supine BP From Baseline in All Participants.
Description: The diastolic supine BP, which is a vital sign parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of treatment-emergent adverse events of potential clinical relevance included abnormal values in body temperature, heart rate, systolic and diastolic blood pressure and respiratory rate that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
mmHg
  Week 4 (N= 69) | 0.1 (8.6)
  Week 8 (N= 61) | -1.3 (8.1)
  Week 12 (N= 58) | -0.9 (7.7)
  Week 16 (N= 53) | 0.3 (8.6)
  Week 20 (N= 44) | -0.0 (9.6)
  Week 24 (N= 45) | 0.4 (9.7)
  Last visit (N= 72) | 0.5 (9.9)

10. Secondary Outcome: Mean Change in Heart Rate From Baseline in All Participants.
Description: The heart rate sitting, which is a vital sign parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of treatment-emergent adverse events of potential clinical relevance included abnormal values in body temperature, heart rate, systolic and diastolic blood pressure and respiratory rate that were identified based on pre-defined criteria. Orthostatic assessments of blood pressure and heart rate were made after the participant was supine for at least 5 minutes and again after the participant was sitting for approximately 2 minutes.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
beats/min
  Week 4 (N= 69) | 1.2 (9.1)
  Week 8 (N= 61) | 1.4 (10.1)
  Week 12 (N= 58) | -1.1 (10.8)
  Week 16 (N= 53) | 4.3 (12.0)
  Week 20 (N= 44) | 3.3 (10.1)
  Week 24 (N= 45) | 0.6 (13.6)
  Last visit (N= 72) | 1.9 (13.0)

11. Secondary Outcome: Mean Change in Systolic BP From Baseline in All Participants.
Description: The systolic sitting BP, which is a vital sign parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of treatment-emergent adverse events of potential clinical relevance included abnormal values in body temperature, heart rate, systolic and diastolic blood pressure and respiratory rate that were identified based on pre-defined criteria. Orthostatic assessments of blood pressure and heart rate were made after the participant was supine for at least 5 minutes and again after the participant was sitting for approximately 2 minutes.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
mmHg
  Week 4 (N= 69) | -0.1 (13.0)
  Week 8 (N= 61) | -0.3 (11.3)
  Week 12 (N= 58) | -0.7 (11.3)
  Week 16 (N= 53) | 1.6 (12.1)
  Week 20 (N= 44) | 1.0 (11.5)
  Week 24 (N= 45) | -0.4 (12.5)
  Last visit (N= 72) | -0.7 (13.4)

12. Secondary Outcome: Mean Change in Diastolic BP From Baseline in All Participants.
Description: The diastolic sitting BP, which is a vital sign parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of treatment-emergent adverse events of potential clinical relevance included abnormal values in body temperature, heart rate, systolic and diastolic blood pressure and respiratory rate that were identified based on pre-defined criteria. Orthostatic assessments of blood pressure and heart rate were made after the participant was supine for at least 5 minutes and again after the participant was sitting for approximately 2 minutes.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
mmHg
  Week 4 (N= 69) | -0.9 (9.7)
  Week 8 (N= 61) | -1.7 (9.4)
  Week 12 (N= 58) | -0.2 (7.9)
  Week 16 (N= 53) | 0.8 (7.8)
  Week 20 (N= 44) | -0.2 (10.0)
  Week 24 (N= 45) | 0.4 (9.8)
  Last visit (N= 72) | 1.4 (10.0)

13. Secondary Outcome: Mean Change in Ventricular Rate From Baseline in All Participants.
Description: The measurement ventricular rate is an ECG parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in heart rate and ECG intervals of PR, RR, QRS, QT, QTcB, QTcN and QTcF that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
Beats/min
  Week 12 (N= 56) | -1.5 (12.0)
  Week 24 (N= 43) | -1.1 (12.3)
  Last visit (N= 70) | -0.1 (13.7)

14. Secondary Outcome: Mean Change in PR Interval From Baseline in All Participants.
Description: The measurement PR interval is an ECG parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in heart rate and ECG intervals of PR, QRS, QT, QTcB, QTcN and QTcF that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
msec
  Week 12 (N= 56) | 3.5 (11.1)
  Week 24 (N= 43) | 0.5 (12.5)
  Last visit (N= 70) | 0.9 (11.6)

15. Secondary Outcome: Mean Change in RR Interval From Baseline in All Participants.
Description: The measurement RR interval is an ECG parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in heart rate and ECG intervals of PR, QRS, QT, QTcB, QTcN and QTcF that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
msec
  Week 12 (N= 56) | 23.7 (140.9)
  Week 24 (N= 43) | 23.3 (152.2)
  Last visit (N= 70) | 8.0 (158.4)

16. Secondary Outcome: Mean Change in QRS Interval From Baseline in All Participants.
Description: The measurement QRS interval is an ECG parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in heart rate and ECG intervals of PR, QRS, QT, QTcB, QTcN and QTcF that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
msec
  Week 12 (N= 56) | -0.1 (5.0)
  Week 24 (N= 43) | 0.4 (5.3)
  Last visit (N= 70) | 0.0 (5.7)

17. Secondary Outcome: Mean Change in QT Interval From Baseline in All Participants.
Description: The measurement QT interval is an ECG parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in heart rate and ECG intervals of PR, RR, QRS, QT, QTcB, QTcN and QTcF that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
msec
  Week 12 (N= 56) | 3.1 (21.5)
  Week 24 (N= 43) | 1.5 (24.9)
  Last visit (N= 70) | 1.0 (25.7)

18. Secondary Outcome: Mean Change in QTcB Interval From Baseline in All Participants.
Description: The measurement QTcB interval is an ECG parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in heart rate and ECG intervals of PR, RR, QRS, QT, QTcB, QTcN and QTcF that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
msec
  Week 12 (N= 56) | -1.6 (20.2)
  Week 24 (N= 43) | -2.4 (19.4)
  Last visit (N= 70) | 0.3 (19.0)

19. Secondary Outcome: Mean Change in QTcF Interval From Baseline in All Participants.
Description: The measurement QTcF interval is an ECG parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in heart rate and ECG intervals of PR, RR, QRS, QT, QTcB, QTcN and QTcF that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
msec
  Week 12 (N= 56) | -0.2 (13.9)
  Week 24 (N= 43) | -1.3 (14.0)
  Last visit (N= 70) | 0.3 (12.9)

20. Secondary Outcome: Mean Change in QTcN Interval From Baseline in All Participants.
Description: The measurement QTcN interval is an ECG parameter were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in heart rate and ECG intervals of PR, RR, QRS, QT, QTcB, QTcN and QTcF that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
msec
  Week 12 (N= 56) | -0.5 (14.7)
  Week 24 (N= 43) | -1.7 (14.3)
  Last visit (N= 70) | 0.3 (13.4)

21. Secondary Outcome: Mean Change in Clinically Relevant Body Weight Changes From Baseline in All Participants.
Description: Clinically relevant body weight changes was one of the primary parameters to measure the safety and tolerability of individual participants. Each participant's body mass index (BMI) kilogram per square meter (kg/m2) were calculated from the screening. Body weight, BMI, and waist circumference changes were evaluated by calculating mean change from Baseline and by tabulating the incidence of ≥7% weight gain or loss.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
Kg
  Week 12 (N= 57) | -0.1 (4.5)
  Week 24 (N= 44) | 1.3 (6.0)
  Last visit (N= 71) | 0.5 (5.8)

22. Secondary Outcome: Mean Change in Clinically Relevant Body Mass Index From Baseline in All Participants.
Description: Clinically relevant body mass index was one of the primary parameters to measure the safety and tolerability of individual participants. Each participant's body mass index (BMI) kilogram per square meter (kg/m2) were calculated from the screening. Body weight, BMI, and waist circumference changes were evaluated by calculating mean change from Baseline and by tabulating the incidence of ≥7% weight gain or loss.
Time Frame: Baseline to last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
Kg/m2
  Week 12 (N= 57) | -0.0 (1.5)
  Week 24 (N= 44) | 0.5 (2.0)
  Last visit (N= 71) | 0.2 (1.9)

23. Secondary Outcome: Mean Change in Clinically Relevant Waist Circumference From Baseline in All Participants.
Description: Clinically relevant waist circumference was one of the primary parameters to measure the safety and tolerability of individual participants. Each participant's body mass index (BMI) kilogram per square meter (kg/m2) were calculated from the screening. Body weight, BMI, and waist circumference changes were evaluated by calculating mean change from Baseline and by tabulating the incidence of ≥7% weight gain or loss.
Time Frame: Baseline to last visit
Population: Safety Sample was analyzed. All enrolled participants who took at least one injection of study medication in the IM depot treatment period. Last visit was defined as the last assessment visit in the treatment phase (scheduled or unscheduled visit). Only Week 24 and last visit data was included.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
cm
  Week 24 (N= 44) | 1.6 (6.6)
  Last visit (N= 64) | 1.3 (6.0)

24. Secondary Outcome: Number of Participants With Clinically Relevant Laboratory Values.
Description: The laboratory values were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal values in serum chemistry, hematology, urinalyses and prolactin tests that were identified based on pre-defined criteria.
Time Frame: Baseline to last visit
Population: All enrolled participants who took at least one injection of study medication in the IM depot treatment period. Last visit was defined as the last assessment visit in the treatment phase (scheduled or unscheduled visit). There were no clinically relevant findings with regard to laboratory values reported in this study.
Measure: Number; unit: participants
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
participants | 0

25. Secondary Outcome: Number of Participants With Clinically Relevant Physical Examination.
Description: The physical examination evaluation was one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in the following body systems: head, ears, eyes, nose, and throat; thorax; abdomen; urogenital; extremities; neurological; and skin and mucosae.
Time Frame: Baseline to last visit
Population: All enrolled participants who took at least one injection of study medication in the IM depot treatment period. Last visit was defined as the last assessment visit in the treatment phase (scheduled or unscheduled visit). None of the abnormalities or findings were noted during physical examination were considered clinically relevant.
Measure: Number; unit: participants
Arm/Group | Aripiprazole IM Depot 400/ 300 mg
Number analyzed (Participants) | 74
participants | 0

ADVERSE EVENTS:
Time Frame: AEs were recorded from the time the ICF was signed until follow-up for safety 14 (±2) days after the last trial visit.
Description: A SAE was any untoward medical occurrence that results in death or was life-threatening or required inpatient hospitalization or prolonged hospitalization. An AE was an exacerbation of an existing problem or any new problem, experienced by a participant when enrolled in a trial, whether or not it was considered drug related by the study physician.
Arm/Group | Aripiprazole IM Depot 400/300 mg
Serious Adverse Events (participants affected / at risk) | 5/74
Other Adverse Events (participants affected / at risk) | 40/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole IM Depot 400/300 mg (N=74)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 2
Schizophrenia (Psychiatric disorders) | 2
Suicidal ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole IM Depot 400/300 mg (N=74)
Weight decreased (Investigations) | 6
Weight increased (Investigations) | 22
Hyperlipidaemia (Metabolism and nutrition disorders) | 4
Akathisia (Nervous system disorders) | 9
Headache (Nervous system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No